CLINICAL TRIAL: NCT04191928
Title: An Exploratory Study of the Pharmacokinetics of Apixaban in Patients Undergoing Pancreaticoduodenectomy
Brief Title: Pharmacokinetics of Apixaban in Patients Undergoing Pancreaticoduodenectomy
Acronym: PAP-UP
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19D.811
Record Dates: First submitted 2019-12-06; First posted 2019-12-10 (Actual); Last update posted 2021-12-23 (Actual); Status verified 2021-12

CONDITIONS: Pancreas Cancer; DVT; Pulmonary Embolism
Keywords: apixaban; pancreaticoduodenectomy; whipple; pharmacokinetic
MeSH Terms: conditions — Pancreatic Neoplasms; Pulmonary Embolism | interventions — apixaban

STUDY DESIGN:
Intervention Model Description: Single-dose pharmacokinetic study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Apixaban dosing (Experimental): Subjects to receive single dose of apixaban
  Interventions: Drug: Apixaban

INTERVENTIONS:
Drug: Apixaban — Apixaban is an orally administered highly selective factor Xa inhibitor, belonging to the class of direct-acting oral anticoagulants (DOAC) along with rivaroxoban and edoxaban. Factor Xa is an essential mediator of the clotting pathway in humans. Apixaban is currently approved by the FDA for treatment of VTE, prophylaxis of DVT in patients undergoing knee and hip replacement surgeries and for reducing the risk of embolic stroke and systemic embolism in patients with nonvalvular atrial fibrillation.
  Other Names: Eliquis

SUMMARY:
Study investigators will examine the absorption characteristics of apixaban, a direct-acting oral anticoagulation, in patients who have underwent a particular kind of surgery (pancreaticoduodenectomy) which involves resection of the duodenum.

DETAILED DESCRIPTION:
This study will examine apixaban pharmacokinetic exposure (AUC(0-24)) and maximum concentration (Cmax) when administered as a single oral dose in patients who have undergone pancreaticoduodenectomy (PD) compared to historical controls. This is a phase one, single dose pharmacokinetic study in stable patients who have undergone pancreaticoduodenectomy. Apixaban is an orally administered highly selective factor Xa inhibitor, belonging to the class of direct-acting oral anticoagulants (DOAC) along with rivaroxoban and edoxaban. Factor Xa is an essential mediator of the clotting pathway in humans. Apixaban is currently approved by the FDA for treatment of VTE, prophylaxis of DVT in patients undergoing knee and hip replacement surgeries and for reducing the risk of embolic stroke and systemic embolism in patients with nonvalvular atrial fibrillation. This study aims to compare the pharmacokinetics and absorption of oral apixaban in patients who have undergone pancreaticoduodenectomy to that of apixaban in historical controls.

ELIGIBILITY:
Inclusion Criteria:

* Be a male or female between ages 18-65 (inclusive) at the screening visit
* May have a history of pharmacologically well-controlled hypertension or non-insulin dependent diabetes
* Have a body mass index (BMI) ≥ 19 and ≤ 33 (inclusive)
* BMI = (weight (kg))/(height (m2))
* Have a history of pancreaticoduodenectomy
* If female, subject can be of childbearing potential and must demonstrate a urine β-hCG level consistent with the non-gravid state at the screening visit and agree to use (and/or have their partner use) an acceptable method of birth control beginning at the screening visit throughout the trial (including washout intervals between treatment periods) and until 2 weeks after the last dose of trial drug in the last treatment period. Acceptable methods of birth control: intrauterine device ("IUD" with or without local hormone release, oral contraceptive pills, diaphragm, cervical cap, spermicides, contraceptive sponge, and /or condoms). Abstinence is an alternative life style and subjects practicing abstinence may be included in the trial.
* Can be of non-childbearing potential which is defined as: a female who is postmenopausal without menses for at least 1 year and an FSH value in the postmenopausal range upon screening evaluation and/or a female who is status post hysterectomy, oophorectomy or tubal ligation.
* Have serum creatinine level < 1.5 mg/dL
* Have a prothrombin time (PT) and activated partial thromboplastin time (PTT) level below the upper limit of normal
* Have platelet count within normal limits
* Be willing to refrain from the use of anticoagulants and antiplatelet medications including aspirin and non-steroidal anti-inflammatory drugs (NSAIDs) during the entire period of study participation
* Be willing to comply with trial restrictions

Exclusion Criteria:

The subject will be excluded from participating in the trial if the subject:

* Has a history of clinically significant medical condition that based upon the judgment of the investigator makes participation inappropriate
* Has a history of a major bleeding event (defined as: (i) symptomatic bleeding in a critical area or organ, such as intracranial, intraspinal, intraocular, retroperitoneal, intra-articular or pericardial, or intramuscular with compartment syndrome, and/or (ii) a fall in hemoglobin level of 2 g/dL or more, or leading to transfusion of two or more units of whole blood or red cells) within 6 months prior to screening visit
* Has had major surgery within 6 months prior to screening visit
* Is actively taking any the following list of medications/supplements and cannot hold these medications for <5 half-lives prior to the study:
* CYP3A4 Moderate/Strong Inhibitors:

Selective Serotonin Reuptake Inhibitors (SSRI) Amiodarone, Dronedarone Diltiazem Cimetidine Aprepitant Protease Inhibitors CYP3A4 Inducers Rifampin Phenytoin Carbemazepine Ritonavir St. John's Wort Enzalutamide Efavirenz Teriflunomide Bosentan Modafinil Mitotane Other Pancreatic Enzyme Replacement (Creon, Pancrelipase, Viokase)

* Has a history of illicit drug abuse within six months prior to screening visit
* Is an active smoker (last exposure <2 weeks prior to study screening)
* Pregnant or lactating
* Consumes greater than 3 glasses of alcoholic beverages (1 glass is approximately equivalent to: beer [354 mL/12 ounces], wine [118 mL/4 ounces], or distilled spirits [29.5 mL/1 ounce]) per day and cannot refrain from alcohol for the duration of the trial
* Has a history of significant multiple and/or severe allergies (e.g. food, drug), or has had an anaphylactic reaction or significant intolerability to prescription or non-prescription drugs or food
* Has known anaphylactic or severe systemic reactions to any components of apixaban or contraindication to the administration of apixaban
* Has moderate or severe hepatic disease or other clinically relevant bleeding risk
* Use of any drugs or products which at the discretion of the investigator would increase bleeding risk
* Is considered inappropriate for participation by the investigator for any reason

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2020-03-03 (Actual); Primary Completion 2020-07-25 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Serum Apixaban Level | 0-24 hours
  Serum apixaban PK level

CONTACTS AND LOCATIONS:
Overall Officials: Walter K Kraft, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University Clinical Research Unit, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No